CLINICAL TRIAL: NCT03280355
Title: The Effects of Singing Training for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Region Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AU_Singing
Record Dates: First submitted 2017-09-01; First posted 2017-09-12 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Randomised controlled trial (RCT); Rehabilitation; Singing Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: Non-pharmacological, intervention based, group randomised (cluster randomised) controlled trial, 2 arms (intervention and active control group)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor (nurse) is masked, primary investigator is masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Singing Training (Experimental): Singing Training as training activity in Pulmonary Rehabilitation: 10 weeks, twice a week for 1 1/2 hour, leading to a total of 20 sessions.
  Interventions: Behavioral: Singing training
- Physical Training (Active Comparator): Physical Training as training activity in Pulmonary Rehabilitation: 10 weeks, twice a week for 1 1/2 hour, leading to a total of 20 sessions.
  Interventions: Behavioral: Physical Training

INTERVENTIONS:
Behavioral: Singing training — Each session will contain technical instruction in order to achieve better respiratory control and primary muscular strength, and with focus on techniques for efficient expiration. Sessions will also focus on musical content and interpretation as well as interaction, the social aspects and joy of singing together.
  Prior to the trial all singing teachers will participate in a 2 days' workshop, where they will be instructed in sufficient methodology and didactics, and will obtain profound knowledge about the disease pathology and related physiology.
  Arms: Singing Training
Behavioral: Physical Training — Physical Training (golden standard training activity in pulmonary rehabilitation) - usual care - is the active comparator in the trial.
  The programme is based on the national guidelines for pulmonary rehabilitation, and consists of supervised warm-ups, aerobic exercises, workout (strength), and breathing exercises.
  Physical Training is conducted by the local physiotherapists in the local health centres.
  Arms: Physical Training

SUMMARY:
Patients with Chronic Obstructive Pulmonary Disease (COPD) experience physiological and psychological complications, such as shortness of breath, anxiety and depression. This has negative influence on their social life, daily activity level and overall quality of life. Patients can participate in a pulmonary rehabilitation program (PR) for the purpose of better managing of the disease and its symptoms and for avoiding future relapses and hospitalisations. However there is a large number of dropouts from PR, and therefore a need for investigation of new activities. Singing training may be one such potential relevant and motivating rehabilitation activity. This study aims to investigate the effects of singing training on both physiological and psychological aspects, and will compare the effects with that of physical training (golden standard in PR). Effects will be investigated in a randomised controlled trial (RCT) with 10 week intervention period. In all the study includes 11 municipalities from around all regions of Denmark, and in all 220 participants.

DETAILED DESCRIPTION:
The number of patients with Chronic Obstructive Pulmonary Disease (COPD) is is rapidly increasing, and the disease is projected to be the third leading cause of death worldwide in 2020. At the present time 320.000 people in Denmark suffer from COPD, though only half of them are diagnosed and hence treated with appropriate medication. Often patients are not diagnosed until the pulmonary function is only 50% and therefore at a severe stage of the disease, where there tends to be a high rate in hospitalisations and recurring exacerbations with increasing symptoms. COPD amounts to 10% of the Danish national health care budget, and Denmark has the highest COPD related mortality rate in the EU.

Besides sufficient medical treatment, patients are offered attendance in pulmonary rehabilitation, since lifestyle changes are crucial in order to prevent disease progression, and for better management of symptoms and higher Quality of Life (QoL). Pulmonary rehabilitation consists of evidence based activities and are based on international and national guidelines. However there is a need for investigation of new motivating and perceived relevant rehabilitation activities due to a large number of drop-outs of the ordinary rehabilitation program.

The study aims to examine the effects of singing training for patients with COPD in relation to physiological as well as psychological aspects. Intervention is singing training, and active control is usual care: Physical training (golden standard and standard part of ordinary pulmonary rehabilitation).

HYPOTHESES:

The main hypothesis of this study is that singing training as activity in pulmonary rehabilitation is non-inferior in relation to effects on specific physiological and specific psychological/psychosocial aspects compared to physical training (control group).

More specifically, the hypotheses are:

1. Singing training leads to a positive rehabilitation process as regards selected physiological parameters as well as selected psychological and psychosocial parameters.
2. Attending the singing training program leads to a more consistent rehabilitation process with higher motivation and less drop outs among the participants than in the control group.

Potential moderators and mediators:

During the project potential mediating and moderating factors will be explored, e.g. including socio-demographic, disease-, lifestyle- and attitude-related characteristics (COPD participants are e.g. characterised by relatively old age and lower socio-economic status). Furthermore, relevant psychological aspects (e.g. in correlation with building and maintaining motivation) will be investigated.

Also baseline attitude towards singing (and physical training), the relationship between the facilitator and participants, and the significance of influence associated with the intervention (e.g. in terms of musical taste) will be taken into consideration.

BACKGROUND:

Physical and psychological effects of COPD:

COPD is a syndrome with a progressive pulmonary obstruction leading to increasingly impaired lung function due to chronic inflammation in the respiratory passages and pulmonary tissue. Living with COPD everyday life is a struggle and often marked by continuous dyspnea, cough and sputum. The patients often suffer from emphysema leading to stiff lungs and insufficient diffusion of oxygen. This again leads to a vicious circle with lack of control of respiratory function, increased hyperinflation and forced, clavicular oriented breathing. Comorbidities such as heart disease, muscle wasting, hypertension and infections are common, which again lead to further complications.

On a psychological level patients are often also affected negatively as a sequela of the disease. E.g. COPD patients tend to suffer from comorbidities such as increased stress and anxiety levels e.g. due to dyspnea. Furthermore patients experience social isolation, financial downfall and generally impaired Quality of Life (QoL). Also activities of daily life are significantly affected by COPD, and the reduced activity again leads to depression and further physical health problems, by which a vicious circle develops. In other words COPD often leads to a severe condition that both physically and psychologically can be very difficult to manage and cope with.

COPD and rehabilitation:

Although the COPD related degeneration of the lungs is irreversible, treatment may slow down further progression, and improve the interrelated physical and psychological consequences of the disease. Besides required medical treatment participants life style change, e.g. smoking cessation, physical training and psychosocial support, are crucial.

According to guidelines from the Danish Government Health Agency patients are encouraged to join an 8-12-wk multidisciplinary rehabilitation program in order to improve physical and mental condition, improve general function and QoL levels, and prevent exacerbations, hospitalisations and early mortality. The overall recommendations are that patients should not only receive clinical control and medical treatment, but should also participate in additional interventions. This is essential in terms of supporting the participants in maintaining (or retrieve) empowerment and self-dependence, also as regards education, work, income, housing and social network.

However, there is a high drop out rate, both due to exacerbations or mortality and to lack of mobility or motivation. Therefore it is of high importance to develop alternative rehabilitation activities that are motivating and are perceived relevant for the participants and that both includes physical training and enables the participants to lead their lives with a higher QoL level. Furthermore, physical and psychological effects of COPD seem to influence each other significantly, suggesting that both areas should be considered in rehabilitation of COPD patients.

There is an unmet need for new types of interventional therapies to help COPD patients. This study aims to investigate singing training as a potential new rehabilitation activity, since singing might lead to a more efficient utilisation of the remaining respiratory function of participants with COPD and improve QoL.

Singing and COPD rehabilitation:

A number of international studies have investigated the effects of singing in relation to COPD patients. The core of singing activity is to learn how to control the respiratory function, including training and coordination of both inspiration and expiration function, focusing on the related primary and secondary musculature. An essential part of the singing training is also focused exercises for posture, relaxation and general body awareness. Moreover, group singing might have a positive impact on the experiences of social interaction, and music in general seems to have an ability to create emotions, and seems to have a positive impact on well-being, anxiety and depression level.

Previous studies differ in methodology (randomized controlled trials, observational studies, qualitative studies and literature reviews), and furthermore sample size and statistical power are not sufficient to conclude on significance and results. Therefore it is of great importance to conduct further and larger trials in order to provide evidence to the field.

In Denmark a number of COPD choirs have been launched, and it seems to have become common-sense that singing is healthy to patients with COPD. The choirs however are launched quite randomly, there is no common methodology on the COPD choirs, and also effects of the choir singing has not yet been investigated. COPD singing therefore has not yet been considered in the national guidelines as a validated rehabilitation activity, however popular among the participants. Therefore the present study is of high relevance, since it aims to provide knowledge and evidence within this field, for the benefit of the large and dramatically growing number of COPD patients.

METHODS:

Study design:

The study is a non-pharmacological two-armed randomized controlled trial with intervention group receiving singing training (ST), and active control group receiving "golden standard": Physical training (PT). Both groups will participate in a 10 weeks' program, 1 1/2 hour, twice a week. Both groups also participate in education activities as part of pulmonary rehabilitation, such as smoking cessation course. Participants randomised to singing training will be offered opportunity to participate in standard physical training post intervention.

ELIGIBILITY:
Inclusion Criteria:

Participants with a clinical diagnosis of COPD and who meet the following criteria are eligible:

1. Recommended for Pulmonary Rehabilitation and minimum mMRC2 level of dyspnea
2. Motivated for participating in the project (and acceptance of randomization)
3. Sufficient mobility to attend PR

Exclusion Criteria:

1. Certain comorbidities (e.g. unstable coronary complications)
2. Severe cognitive disabilities (e.g. dementia)
3. Inability to speak or understand Danish

No previous singing experience or musical competence is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
6 Minutes Walk Distance (6MWD) | 12 weeks (+/- 2 weeks)
  Meters

SECONDARY OUTCOMES:
Pedometer | 12 weeks (+/- 2 weeks)
  Number of steps (worn for 1 week (7 days) at baseline and post intervention)
St. George's Respiratory Questionnaire (SGRQ) | 12 weeks (+/- 2 weeks)
  Quality of Life-questionnaire (self-reported)
Forced Expiratory Volume Predicted (FEV1%) | 12 weeks (+/- 2 weeks)
  The FEV1% is the FEV1 divided by the FVC (Forced Vital Capacity) times 100: FEV1%=FEV1/VC X100
Breath Hold Test | 12 weeks (+/- 2 weeks)
  Number of seconds (from max inspiration)
Single-breath Count | 12 weeks (+/- 2 weeks)
  Numbers counted (beats per minute=60) (from max inspiration)
Compliance | 10 weeks
  Self-produced excel sheet with registration each time of each participant's attendance or absence (with or without cause). Registered continuously during intervention period.
Musical Ear Test (MET) | 12 weeks (+/- 2 weeks)
  Test for musical competence: 104 trials on which participants judge whether two short musical phrases (melody/rhythm) are identical or not

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Bodtger, MD PhD, Principal Investigator — Region Zealand; Peter Vuust, Professor, Study Director — Aarhus Univeristy
Locations (11):
- Denmark (11):
  - Rudersdal Health Centre, Birkerød
  - Helsingor Health Centre, Elsinore
  - Fakse Health Centre, Fakse
  - Vesthimmerland Health Centre, Farsø
  - Hedensted Health Centre, Hedensted
  - Ikast-Brande Health Centre, Ikast
  - Lemvig Health Centre, Lemvig
  - Lolland Health Centre, Maribo
  - Silkeborg Health Centre, Silkeborg
  - Slagelse Health Centre, Slagelse
  - Vordingborg Health Centre, Vordingborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaasgaard M, Rasmussen DB, Andreasson KH, Hilberg O, Lokke A, Vuust P, Bodtger U. Use of Singing for Lung Health as an alternative training modality within pulmonary rehabilitation for COPD: a randomised controlled trial. Eur Respir J. 2022 May 19;59(5):2101142. doi: 10.1183/13993003.01142-2021. Print 2022 May. PMID 34625480
- [Derived] Kaasgaard M, Andersen IC, Rasmussen DB, Hilberg O, Lokke A, Vuust P, Bodtger U. Heterogeneity in Danish lung choirs and their singing leaders: delivery, approach, and experiences: a survey-based study. BMJ Open. 2020 Nov 30;10(11):e041700. doi: 10.1136/bmjopen-2020-041700. PMID 33257493

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT03280355/SAP_000.pdf